CLINICAL TRIAL: NCT02191371
Title: Effect of Anesthetics on Oxygenation and Microcirculation During One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PaO2 & StO2 in OLV
Record Dates: First submitted 2014-07-07; First posted 2014-07-16 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2014-08

CONDITIONS: Mechanical Ventilation Complication
Keywords: oxygenation; microcirculation; one-lung ventilation; thoracic surgery
MeSH Terms: interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol (Experimental): Propofol is used as a maintenance anesthetic to patients in the propofol group. Intervention: propofol infusion by target-controlled infusion for maintaining anesthesia propofol (Fresofol MCT 2%) target effect site concentration: 4~5 mcg/ml, during general anesthesia
  Interventions: Drug: propofol
- desflurane (Experimental): Desflurane is used as a maintenance anesthetic to patients in the desflurane group.
  Intervention: Desflurane administration for maintaining anesthesia desflurane (Suprane) inhalation as 6~8 vol% during general anesthesia
  Interventions: Drug: desflurane

INTERVENTIONS:
Drug: propofol — Patients are randomized to receive intravenous anesthetic (propofol) or inhalational anesthetic (desflurane) as a maintenance anesthetic.
  Other Names: propofol (Fresofol(R)2 MCT 2%, Fresenius Kabi)
  Arms: propofol
Drug: desflurane — Patients are randomized to receive intravenous anesthetic (propofol) or inhalational anesthetic (desflurane) as a maintenance anesthetic.
  Other Names: desflurane (Suprane(R), Baxter Healthcare)
  Arms: desflurane

SUMMARY:
One-lung ventilation during thoracic surgery may affect systemic oxygenation and peripheral microcirculation by hypoxic pulmonary vasoconstriction. Both intravenous and inhalational anesthetics can be used during one-lung ventilation. However, there is still a controversy which anesthetic would be more appropriate during one-lung ventilation in the perspective of oxygenation and microcirculation. The investigators hypothesized that intravenous and inhalational anesthetics may affect oxygenation and microcirculation differently during one-lung ventilation.

DETAILED DESCRIPTION:
Patients undergoing thoracic surgery including one-lung ventilation will be randomized to receive intravenous (propofol) or inhalational (desflurane) anesthetic.

Systemic oxygenation can be evaluated by measuring partial pressure of oxygen in arterial blood analysis. Microcirculatory parameters can be obtained from vascular occlusion test. Among those parameters, recovery slope during vascular occlusion test is known to reflect recruitment of microvasculature in response to hypoxic or ischemic insult. In this study, we will compare arterial partial pressure of oxygen and recovery slope during one-lung ventilation between propofol and desflurane group.

ELIGIBILITY:
Inclusion Criteria:

* undergoing thoracic surgery including one-lung ventilation

Exclusion Criteria:

* refuse to enroll
* BMI over 30 kg/m(2)
* severe obstructive or restrictive lung disease
* preoperative supplemental oxygen, intubated, or mechanical ventilatory support
* preoperative arterial partial pressure of oxygen < 60 mmHg
* pregnancy
* history of coronary artery disease
* preoperative continuous infusion of vasopressor or inotropes
* cannot undergo vascular occlusion test: anatomical abnormality of both arms, severe peripheral vascular disease, presence of A-V fistula

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
arterial partial pressure of oxygen | 30 min after one-lung ventilation
  Primary outcome is arterial partial pressure of oxygen 30 min after one-lung ventilation during thoracic surgery in propofol and desflurane groups.

SECONDARY OUTCOMES:
recovery slope | 30 min after one-lung ventilation
  Secondary outcome is recovery slope measured by vascular occlusion test 30 min after one-lung ventilation during thoracic surgery in propofol and desflurane groups.

OTHER OUTCOMES:
blood pressure | 30 min after one-lung ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho YJ, Kim TK, Hong DM, Seo JH, Bahk JH, Jeon Y. Effect of desflurane-remifentanil vs. Propofol-remifentanil anesthesia on arterial oxygenation during one-lung ventilation for thoracoscopic surgery: a prospective randomized trial. BMC Anesthesiol. 2017 Jan 18;17(1):9. doi: 10.1186/s12871-017-0302-x. PMID 28100177